CLINICAL TRIAL: NCT04144413
Title: A Phase IIIb, Prospective, Interventional, Multicentre, 3-year Study to Explore the Long-term Evolution of Sign and Symptoms, and Occurence of Complications in Dry Eye Patients With Severe Keratitis Receiving Ikervis® (1mg/mL Ciclosporin)
Brief Title: 3-year Study in Dry Eye Disease Patients With Severe Keratitis Receiving Ikervis® (1mg/mL Ciclosporin)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NVG14L127
Record Dates: First submitted 2019-10-25; First posted 2019-10-30 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Dry Eye Disease With Severe Keratitis

STUDY DESIGN:
Intervention Model Description: In order to assess the response to IKERVIS® for DED patients with severe keratitis, after 12-month IKERVIS® (once daily) treatment, patients who have shown a marked improvement at Month 12 (as defined below) will be randomised to receive IKERVIS® or Vehicle (ration 3:2) in double-masked fashion.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Period 1 Open-label Ikervis (Experimental): Period 1 for all patients: IKERVIS® (1mg/ml CsA). Instillation of one drop in each affected eye, once daily at bedtime. From Baseline for the first 12 months of treatment.
  Interventions: Drug: Open-label Ikervis
- Period 2 Masked Ikervis (Experimental): Period 2 for markedly improved patients at Month 12 only, and double-masked fashion.
  IKERVIS® (1mg/ml CsA). Instillation of one drop in each affected eye, once daily at bedtime. From Month 12 to Month 36.
  Interventions: Drug: Masked Ikervis
- Period 2 Masked Vehicle (Other): Other: Vehicle Comparator. Period 2 for markedly improved patients at Month 12 only, and double-masked fashion.
  Vehicle. Instillation of one drop in each affected eye, once daily at bedtime. From Month 12 to Month 36.
  Interventions: Other: Vehicle Comparator: Masked Vehicle

INTERVENTIONS:
Drug: Open-label Ikervis — NOVA22007, IKERVIS® is a sterile, ophthalmic cationic oil-in-water emulsion containing 1mg/ml CsA.
  Arms: Period 1 Open-label Ikervis
Drug: Masked Ikervis — NOVA22007, IKERVIS® is a sterile, ophthalmic cationic oil-in-water emulsion containing 1mg/ml CsA.
  Arms: Period 2 Masked Ikervis
Other: Vehicle Comparator: Masked Vehicle — Vehicle of IKERVIS® - sterile, ophthalmic cationic oil-in-water emulsion containing no active substance.
  Arms: Period 2 Masked Vehicle

SUMMARY:
The proposed 36-month Post Approval Efficacy Study (PAES) is a prospective, interventional, multicentre study to explore the long-term evolution of signs and symptoms, and occurrence of complications in Dry Eye Disease (DED) patients with severe keratitis receiving Ikervis® (1mg/mL ciclosporin) eye drops administered once daily

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the patient is capable of understanding and complying with protocol requirements.
2. The patient has signed and dated a written informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Male or female patient is aged 18 years or above.
4. At least 4 weeks of use of tear substitutes prior to the Baseline Visit
5. DED patients with severe keratitis defined as the following:

   * CFS score of 3, 4 or 5 on the modified Oxford scale in at least one eye at Baseline Visits, AND
   * Schirmer test without anaesthesia scored <10 mm/5min in the same eye at Baseline Visit, AND
   * At least two moderate to very severe symptoms of dry eye disease with a score ≥2 (severity graded on a 0 to 4 grade scale), among the following symptoms: burning/stinging, foreign body sensation, eye dryness, eye pain and blurred/poor vision at Baseline Visit.
6. Patient must be willing and able to undergo and return for scheduled study-related examinations.

Exclusion Criteria:

1. Active herpes keratitis or history of ocular herpes.
2. History of ocular trauma or ocular infection (viral, bacterial, fungal, protozoal) within 90 days before the Baseline Visit.
3. Any ocular diseases other than DED requiring topical ocular treatment during the course of the study. Patients taking preservative-free IOP lowering medications are eligible for study enrolment.
4. Concurrent ocular allergy (including seasonal conjunctivitis) or chronic conjunctivitis other than dry eye.
5. Anticipated use of temporary punctal plugs during the study. Patients with punctal plugs placed prior to the Baseline Visit are eligible for enrolment; however, punctal plugs must remain in place during the study.
6. Best corrected distance visual acuity (BCDVA) score ≤ 20/200 Snellen in each eye.
7. Presence or history of any systemic or ocular disorder, condition or disease that could possibly interfere with the conduct of the required study procedures or the interpretation of study results or judged by the investigator to be incompatible with the study (e.g., diabetes with glycemia out of range, thyroid malfunction, uncontrolled autoimmune disease, current systemic infections, ocular infection…).
8. Known hypersensitivity to one of the components of the study or procedural medications (e.g., fluorescein, etc.).
9. History of ophthalmic malignancy
10. History of malignancy (other than ophthalmic) in the last 5 years.
11. Anticipated change during course of the study in the dose of systemic medications that could affect a dry eye condition [mainly, estrogen-progesterone or other estrogen derivatives (only allowed for post-menopausal women), pilocarpine, isotretinoine, tetracycline, antihistamines, tricyclic antidepressants, anxiolytics, antimuscarinics, beta-blocking agents, phenothiazines, omega-3, systemic corticosteroids]. These treatments are allowed during the study provided they remain stable throughout the course of the study.
12. Use of topical ciclosporin in the past 3 months prior to Baseline visit.
13. Any change in systemic immunosuppressant drugs within 30 days before the Baseline Visit or anticipated change during the course of the study.
14. Pregnancy or lactation at the Baseline Visit.
15. Women of childbearing potential not using a medically acceptable, highly effective method of birth control (such as hormonal implants, injectable or oral contraceptives together with condoms, some intrauterine devices, sexual abstinence or vasectomised partner) from the Baseline Visit throughout the conduct of the study treatment periods and up to 2 weeks after the study end. Post-menopausal women (two years without menstruation) do not need to use any method of birth control.
16. Participation in a clinical trial with an investigational substance within the past 30 days prior to Baseline Visit.
17. Participation in another clinical study at the same time as the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Sébastien GARRIGUE, PhD, Study Chair — Santen SAS
Locations (45):
- Czechia (8):
  - Fakultni Nemocnice Ostrava, Oční Klinika, Ostrava, Moravskoslezský kraj
  - University Hospital Hradec Kralove, Hradec Králové, Nový Hradec Králové
  - Ocni klinika OFTEX, Pardubice, Pardubický kraj
  - MEDOKO s.r.o., Prague, Prague
  - Axon clinical s.r.o., Prague, Prague
  - Fakultní Nemocnice Brno, Brno, South Moravian
  - Nemocnice Teplice, Ocni Oddeleni, Teplice, Ústecký kraj
  - Masarykova nemocnice, Ocni oddeleni, Ústí nad Labem, Ústecký kraj
- France (4):
  - Hospices Civils de Lyon - Hopital de la Croix-Rousse, Lyon, Auvergne-Rhône-Alpes
  - Hopitaux Universitaires Paris-Sud - Hopital Bicetre, Le Kremlin-Bicêtre, Île-de-France Region
  - Hôpital des Quinze-Vingts, Paris, Île-de-France Region
  - Hopitaux Universitaires Paris Nord Val de Seine - Hopital Bichat - Claude Bernard, Paris, Île-de-France Region
- Italy (7):
  - Universita degli Studi di Milano - Clinica Oculistica I, Milan, Lombardy
  - Universita degli Studi di Milano - Ospedale San Giuseppe - Clinica Oculistica (University Eye Clinic), Milan, Lombardy
  - ASST Santi Paolo e Carlo - Ospedale San Paolo Polo Universitario - Clinica Oculistica III, Milan, Lombardy
  - Polo Universita degli Studi di Milano - Ospedale Luigi Sacco - Clinica Oculistica (Eye Clinic), Milan, Lombardy
  - Universita degli Studi di Pavia - Fondazione IRCCS Policlinico San Matteo - Clinica Oculistic, Pavia, Lombardy
  - Azienda Ospedaliera Universitaria Policlinico Gaetano Martino - Messina, Messina, Sicily
  - Universita degli Studi di Padova - Azienda Ospedaliera di Padova - Clinica Oculistica, Padua, Veneto
- Poland (6):
  - Niepubliczny Zaklad Opieki Zdrowotnej Oko-Laser, Krakow, Lesser Poland Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 Klinika Diagnostyki i Mikrochirurgii Jaskry Oddział Okulistyki, Lublin, Lublin Voivodeship
  - Gabinet Okulistyczny Prof. Edward Wylęgała, Katowice, Silesian Voivodeship
  - Uniwersyteckie Centrum Kliniczne Śląskiego Uniwersytetu Medycznego w Katowicach, Katowice, Silesian Voivodeship
  - Retina Szpital Okulistyczny, Warsaw, Warszawskie
  - Uniwersytecki Szpital Kiliniczny IM. Jana Milkulicza-Radeckiego we Wroclawiu, Wroclaw, Wrocławiu
- Russia (9):
  - Federal State Institution Intersectoral Research and Technology Complex Eye microsurgery n.a. academician S.N. Fyodorov - Cheboksary, Cheboksary, Chuvashskaya Respublika
  - Ivanovo Regional Clinical Hospital, Ivanov, Ivanovo Oblast
  - State Budget Educational Institution of High Professional Education Moscow State Medical Stomatology University named after A.I.Evdokimov of MoH of RF, Moscow, Moscow
  - NMRC ISTC Eye Microsurgery n. a. Fyodorov - Moscow, Moscow, Moscow
  - Saint Petersburg State Pediatric Medical University, Saint Petersburg, Sankt-Peterburg
  - First Saint Petersburg State Medical University named after academician I.P. Pavlov, Saint Petersburg, Sankt-Peterburg
  - FSBI The Academician S.N. Fyodorov IRTC Eye Microsurgery of the Minzdrava - Novosibirsk, Novosibirsk
  - GBOU VPO Omsk State Medical Academy, Ophthalmology Department, Omsk
  - Saratov Railway Clinic, Saratov
- Spain (7):
  - Cartujavision Oftalmologia, Seville, Andalusia
  - Hospital Clinico Universitario Lozano Blesa de Zaragoza, Zaragoza, Aragon
  - Hospital Universitario Donostia, Oftalmalogia, Donostia / San Sebastian, Basque Country
  - Institut Catala de Retina, Barcelona, Catalonia
  - Centro de Oftalmología Barraquer, Barcelona, Catalonia
  - Hospital Clinic de Barcelona (Hospital Clinic i Provincial), Barcelona, Catalonia
  - Fundación Oftalmológica del Mediterráneo, Valencia
- Turkey (Türkiye) (4):
  - Bayındır Kavaklidere Hospital Ophthalmology department, Ankara, Anatolia
  - Ankara Üniversitesi Tıp Fakültesi Göz Hastalıkları Anabilim Dalı Vehbi Koç Göz Hastanesi, Mamak, Ankara
  - Ege Universitesi Tip Fakultesi Hastanesi Goz Hastaliklari Anabilim Dali, Bornova, İzmir
  - Selcuk University School of Medicine Ophthalmology department, Konya, Selcuklu

RESULTS

PARTICIPANT FLOW:
Groups:
- Period 1 Open-Label Treatment Ikervis: Period 1 for all patients: IKERVIS® (1mg/ml CsA). Instillation of one drop in each affected eye, once daily at bedtime. From Baseline for the first 12 months of treatment.
  Open-Label Ikervis: NOVA22007, IKERVIS® is a sterile, ophthalmic cationic oil-in-water emulsion containing 1mg/ml CsA.
- Period 2 Masked Treatment Ikervis: Period 2 for markedly improved patients at Month 12 only, and double-masked fashion.
  IKERVIS® (1mg/ml CsA). Instillation of one drop in each affected eye, once daily at bedtime. From Month 12 to Month 36.
  Masked Ikervis: NOVA22007, IKERVIS® is a sterile, ophthalmic cationic oil-in-water emulsion containing 1mg/ml CsA.
- Period 2 Masked Treatment Vehicle: Other: Vehicle Comparator. Period 2 for markedly improved patients at Month 12 only, and double-masked fashion.
  Vehicle: Instillation of one drop in each affected eye, once daily at bedtime. From Month 12 to Month 36.
  Vehicle Comparator is Masked Vehicle: Vehicle of IKERVIS® - sterile, ophthalmic cationic oil-in-water emulsion containing no active substance.
Period: Period 1: Open-Label Treatment Phase
Arm/Group | Period 1 Open-Label Treatment Ikervis | Period 2 Masked Treatment Ikervis | Period 2 Masked Treatment Vehicle
Started | 350 | 0 | 0
Completed | 288 (62 participants exited the study prematurely and 288 completed the Open-Label Treatment Period 1 at Month 12.) | 0 | 0
Not Completed | 62 | 0 | 0
Period: Period 2: Masked Treatment Phase
Arm/Group | Period 1 Open-Label Treatment Ikervis | Period 2 Masked Treatment Ikervis | Period 2 Masked Treatment Vehicle
Started | 0 | 148 (Out of the 288 completed participants at Month 12 in Period 1, 245 subjects were randomized to 2 treatment groups in a 3:2 ratio (n = 148 to IKERVIS® and n = 97 to vehicle)) | 97 (Out of the 288 completed participants at Month 12 in Period 1, 245 subjects were randomized to 2 treatment groups in a 3:2 ratio (n = 148 to IKERVIS® and n = 97 to vehicle))
Completed | 0 | 137 (22 participants exited the study prematurely and 223 completed the Double Masked Treatment Period 2 at Month 36.) | 86 (22 participants exited the study prematurely and 223 completed the Double Masked Treatment Period 2 at Month 36.)
Not Completed | 0 | 11 | 11

BASELINE CHARACTERISTICS:
Arm/Group | Period 1 Open-Label Treatment Ikervis
Number analyzed (Participants) | 350
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 209
  >=65 years | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (13.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 302
  Male | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 51
  Not Hispanic or Latino | 298
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 11
  Black or African American | 1
  White | 331
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 10
  Czechia | 65
  Poland | 83
  Italy | 57
  Russia | 61
  Spain | 74

OUTCOME MEASURES:

1. Primary Outcome: The Correlation Between Mean Change From Baseline in Corneal Fluorescein Staining (CFS) Score and Symptom Assessment iN Dry Eye (SANDE) Symptoms Score at Each Visit.
Description: For analysis, SCC (Spearman Correlation Coefficient) and its 95% Confidence Interval were calculated for the correlation analysis between change from baseline in CFS (Corneal Fluorescein Staining) score at visit X and SANDE (Symptom Assessment iN Dry Eye) symptoms score using the FAS (Full Analysis Set) Period 1 Population.
Time Frame: Months 3, 6, 9, and 12
Population: Full Analysis Set (FAS). The number of analyzed data are participants evaluable for the outcome measure at Months 3, 6, 9, and 12.
  Comment3: Overall Number of Participants analyzed were 336 who received at least one dose of the study medication and had at least one post-baseline sign or symptom assessment of the study eye during Period 1. However, the discrepancy between each specific time-frame is due to missing data or patients withdrawn. These statistical methods were defined in a SAP.
Measure: Mean (95% Confidence Interval); unit: Spearman Correlation Coefficient
Arm/Group | Period 1 Open-Label Treatment Ikervis
Number analyzed (Participants) | 336
Spearman Correlation Coefficient
  Month 3 / Month 3: number analyzed (Participants) | 318
  Month 3 / Month 3 | 0.169 [0.060 to 0.274]
  Month 3 / Month 6: number analyzed (Participants) | 272
  Month 3 / Month 6 | 0.245 [0.130 to 0.353]
  Month 3 / Month 9: number analyzed (Participants) | 274
  Month 3 / Month 9 | 0.274 [0.160 to 0.380]
  Month 3 / Month 12: number analyzed (Participants) | 275
  Month 3 / Month 12 | 0.178 [0.060 to 0.290]
  Month 6 / Month 6: number analyzed (Participants) | 275
  Month 6 / Month 6 | 0.258 [0.144 to 0.365]
  Month 6 / Month 9: number analyzed (Participants) | 262
  Month 6 / Month 9 | 0.322 [0.209 to 0.426]
  Month 6 / Month 12: number analyzed (Participants) | 263
  Month 6 / Month 12 | 0.274 [0.158 to 0.382]
  Month 9 / Month 9: number analyzed (Participants) | 274
  Month 9 / Month 9 | 0.343 [0.234 to 0.444]
  Month 9 / Month 12: number analyzed (Participants) | 268
  Month 9 / Month 12 | 0.332 [0.221 to 0.434]
  Month 12 / Month 12: number analyzed (Participants) | 288
  Month 12 / Month 12 | 0.266 [0.155 to 0.370]

2. Secondary Outcome: Corneal Fluorescein Staining (CFS) Score and Change From Baseline by Visit
Description: Period 1 is Baseline to Month 12 included. CFS is Corneal Fluorescein Score. Staining using fluorescein was graded using the modified Oxford scale (7-point ordinal scale, score 0, 0.5, and 1 to 5 per area [cornea + nasal and temporal conjunctiva]) for cornea and conjunctiva separately. On this modified scale, the score 0 corresponds to no staining dots and the score 0.5 corresponds to one staining dot per area.
  A CFS grade of 0 represents complete corneal clearing.
Time Frame: Baseline, Months 3, 6, 9 and 12
Population: Full Analysis Set (FAS). The number of analyzed data are participants evaluable for the outcome measure at Baseline, Months 3, 6, 9, and 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Period 1 Open-Label Treatment Ikervis
Number analyzed (Participants) | 336
score on a scale
  Observed Baseline | 3.62 (0.667)
  Observed Month 3: number analyzed (Participants) | 321
  Observed Month 3 | 2.24 (1.072)
  Month 3 change from baseline: number analyzed (Participants) | 321
  Month 3 change from baseline | -1.38 (0.995)
  Observed Month 6: number analyzed (Participants) | 276
  Observed Month 6 | 1.72 (1.137)
  Month 6 change from baseline: number analyzed (Participants) | 276
  Month 6 change from baseline | -1.91 (1.143)
  Observed Month 9: number analyzed (Participants) | 274
  Observed Month 9 | 1.42 (1.094)
  Month 9 change from baseline: number analyzed (Participants) | 274
  Month 9 change from baseline | -2.20 (1.123)
  Observed Month 12: number analyzed (Participants) | 288
  Observed Month 12 | 1.14 (1.008)
  Month 12 change from baseline: number analyzed (Participants) | 288
  Month 12 change from baseline | -2.49 (0.981)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent and were followed to resolution or until the subject's participation in the study ended for both Period 1 (Open-Label Treatment Period) at Month 12 and Period 2 (Double Masked Treatment Period) at Month 36.
Description: Other Adverse Events data is a summary observed at a rate of 0% or higher by System Organ Class and Preferred Term for both the Open-Label and Double Masked Periods. The summary of other adverse events in Open Label Treatment Period and Double Masked Treatment Period are independently summarized.
Groups:
- Period 1 Open-Label Treatment Ikervis: Period 1 for all patients: IKERVIS® (1mg/ml CsA). Instillation of one drop in each affected eye, once daily at bedtime. From Baseline for the first 12 months of treatment.
  Open-Label Ikervis: NOVA22007, IKERVIS® is a sterile, ophthalmic cationic oil-in-water emulsion containing 1mg/ml CsA.
  Comment 4: The number of enrolled participants were 350, however, 344 participants received at least 1 dose of study medication and were included in the Safety Population Entire Study analysis. Participants who didn't receive study medicaiton were not included in the safety population. These statistical methods were defined in a pre-created statistical analysis plan.
Arm/Group | Period 1 Open-Label Treatment Ikervis | Period 2 Masked Treatment Ikervis | Period 2 Masked Treatment Vehicle
All-Cause Mortality (participants affected / at risk) | 1/344 | 0/148 | 0/97
Serious Adverse Events (participants affected / at risk) | 15/344 | 12/148 | 9/97
Other Adverse Events (participants affected / at risk) | 138/344 | 58/148 | 39/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1 Open-Label Treatment Ikervis (N=344) | Period 2 Masked Treatment Ikervis (N=148) | Period 2 Masked Treatment Vehicle (N=97)
COVID-19 (Infections and infestations) | 4 | 2 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
Brain Stem Stroke (Nervous system disorders) | 1 | 0 | 0
Superior sagittal sinus thrombosis (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0
Posterior capsule opacification (Eye disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Sialoadenitis (Infections and infestations) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Genital prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
Coronary artery bypass (Surgical and medical procedures) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1 Open-Label Treatment Ikervis (N=344) | Period 2 Masked Treatment Ikervis (N=148) | Period 2 Masked Treatment Vehicle (N=97)
Eye irritation (Eye disorders) | 26 (28) | 4 (4) | 0 (0)
Eye pain (Eye disorders) | 16 (18) | 0 (0) | 2 (2)
Dry Eye (Eye disorders) | 15 (15) | 3 (3) | 5 (5)
Eye pruritus (Eye disorders) | 12 (12) | 3 (4) | 1 (1)
Ocular hyperaemia (Eye disorders) | 11 (11) | 3 (3) | 0 (0)
Visual acuity reduced (Eye disorders) | 4 (5) | 3 (4) | 3 (3)
Conjunctival hyperaemia (Eye disorders) | 4 (4) | 1 (1) | 2 (2)
Lacrimation increased (Eye disorders) | 3 (4) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 4 (4) | 3 (3) | 1 (1)
Abnormal sensation in eye (Eye disorders) | 3 (3) | 1 (1) | 1 (1)
Chalazion (Eye disorders) | 3 (3) | 1 (2) | 2 (2)
Conjunctival oedema (Eye disorders) | 3 (3) | 1 (1) | 1 (1)
Ocular discomfort (Eye disorders) | 3 (3) | 1 (1) | 0 (0)
Blepharospasm (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Corneal leukoma (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Corneal oedema (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 2 (2) | 1 (1) | 1 (1)
Eyelids pruritus (Eye disorders) | 2 (2) | 0 (0) | 1 (1)
Foreign body sensation in eyes (Eye disorders) | 2 (2) | 3 (3) | 2 (2)
Keratitis (Eye disorders) | 2 (2) | 1 (1) | 2 (2)
Lenticular opacities (Eye disorders) | 2 (2) | 2 (2) | 0 (0)
Meibomian gland dysfunction (Eye disorders) | 2 (2) | 1 (1) | 1 (1)
Noninfective conjunctivitis (Eye disorders) | 1 (2) | 0 (0) | 1 (1)
Noninfective conjunctivitis (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 5 (5) | 3 (5)
Cataract (Eye disorders) | 1 (1) | 5 (6) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dacryolith (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatochalasis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema eyelids (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema of eyelid (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
Lacrimation disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ocular hypertension (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Pinguecula (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 8 (8) | 10 (11) | 5 (5)
Conjunctivitis (Infections and infestations) | 4 (5) | 3 (4) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (4) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 3 (3) | 1 (3) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (2) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Asymptomatic COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Eye infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Eyelid infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Instillation site pain (General disorders) | 3 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Instillation site paraesthesia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Product intolerance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Facial neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine with aura (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Foreign body in eye (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Soft tissue foreign body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Varicose ulceration (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Blood cholesterol (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Adnexa uteri cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 2 (2) | 3 (3) | 1 (1)
Posterior capsule opacification (Eye disorders) | 0 (0) | 2 (2) | 2 (2)
Corneal degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Episcleritis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye allergy (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Meibomianitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vitreoretinal traction syndrome (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eyelash discolouration (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Macular cyst (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Meibomian gland discharge (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Trichiasis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes ophthalmic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lyme disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Borrelia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dandruff (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Lens extraction (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hip surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Foot operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 1 (1) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Vital dye staining cornea present (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Eyelid haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vocal cord inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Lacrimal disorder (Eye disorders) | 0 (0) | 2 (3) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT04144413/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT04144413/SAP_001.pdf